CLINICAL TRIAL: NCT02714491
Title: Effects of Auditory Stimulation During Verticalization With Erigo in Patients With Disorder of Consciousness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Principal Investigator, Ilaria Zivi, MD, Ospedale Generale Di Zona Moriggia-Pelascini
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Erigo.stim
Record Dates: First submitted 2016-03-10; First posted 2016-03-21 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Consciousness Disorders
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Music (Active Comparator): Erigo + Music: During each stepping verticalization session the patient receives auditory stimulation (earphones) with previously preferred music
  Interventions: Other: Erigo + Music
- Metronome (Active Comparator): Erigo + Metronome: During each stepping verticalization session the patient receives auditory stimulation (earphones) with a metronome (rhythmic with the stepping movement)
  Interventions: Other: Erigo + Metronome
- Silence (Active Comparator): Erigo + Silence: During each stepping verticalization session the patient does note receive any auditory stimulation.
  Interventions: Other: Erigo + Silence

INTERVENTIONS:
Other: Erigo + Music — The patients receive daily conventional physiotherapy + fifteen 30-minutes stepping verticalization sessions with "Erigo" (3/week for 5 consecutive weeks) and musical stimulation.
  Arms: Music
Other: Erigo + Metronome — The patients receive daily conventional physiotherapy + fifteen 30-minutes stepping verticalization sessions with "Erigo" (3/week for 5 consecutive weeks) and metronome stimulation.
  Arms: Metronome
Other: Erigo + Silence — The patients receive daily conventional physiotherapy + fifteen 30-minutes stepping verticalization sessions with "Erigo" (3/week for 5 consecutive weeks), without auditory stimulation.
  Arms: Silence

SUMMARY:
Aim of the study is to define if the auditory stimulation during stepping verticalization sessions with "Erigo" is able to modify the cerebral electric activity or improve consciousness in patients affected by vegetative state or minimally conscious state.

ELIGIBILITY:
Inclusion Criteria:

* Vegetative State or Minimally Conscious State diagnosis
* >3 months from acute brain injury

Exclusion Criteria:

* No clinical stability
* Sepsis
* Orthopaedic contraindications for verticalization
* Deep Vein Thrombosis
* weight >130 Kg
* height >210 cm

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
change in Coma Recovery Scale revised score | 0 and 35 days

SECONDARY OUTCOMES:
change in Levels of Cognitive Functioning score | 0 and 35 days
change in Disability Rating Scale score | 0 and 35 days
change in quantitative EEG parameters | 0 and 35 days
change in Glasgow Coma Scale score | 0 and 35 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Generale di Zona Moriggia Pelascini, Gravedona Ed Uniti, CO, Italy